CLINICAL TRIAL: NCT01070667
Title: Dronedarone in Pacemaker Patients With Paroxysmal Atrial Fibrillation
Brief Title: Dronedarone in Pacemakers Patients With Paroxysmal Atrial Fibrillation
Acronym: DROPPAF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastbourne General Hospital (Other)
Responsible Party: Dr AN Sulke, East Sussex NHS Trust
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DROPPAF V2.1
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: PAF; AF; Dronedarone; AF Burden; AFB; PPM; Permanent Pacemaker; Atrial Fibrillation Burden in Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dronedarone (Experimental): Patients will receive 400 mg of dronedarone per day for 3 months.
  Interventions: Drug: Dronedarone
- Placebo (Placebo Comparator): Patients will receive a placebo tablet once per day for 3 months. AF burden and other parameters described will be monitored from the participants permanent pacemaker. Participants will also be asked to fill out symptom diaries and questionaires.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronedarone — 400mg orally once per day for 3 months
  Other Names: Multaq
  Arms: Dronedarone
Drug: Placebo — 1 tablet once per day for 3 months. The tablet will appear identical to the active dronedarone tablet.
  Arms: Placebo

SUMMARY:
The purpose of this study is to accurately investigate the efficacy of dronedarone in maintaining sinus rhythm and decreasing AFB in patients with paroxysmal atrial fibrillation as compared with placebo. This has never previously been performed using pacemaker Holter monitoring which provides detailed information of atrial arrhythmia patterns the entire study period. Additionally detailed patient symptom self assessment and questionnaires will be collected. The study design will be double blinded crossover with each phase lasting 3 months.

DETAILED DESCRIPTION:
The study is planned to commence in March 2010 after obtaining Ethics Committee approval. Patients will be randomised to a three month course of dronedarone or placebo. 1:1 double blinded randomisation will be undertaken. At three months, after a one week washout period, the patients will cross-over treatment groups. To achieve a power of 0.8 with a type one error rate 5% detecting a relative difference of 10% primary outcomes the study will require 42 patients. 50 patients in total will be enrolled in the study. The study will take place at Eastbourne District General Hospital. The study duration per patient is 7 months. The overall study duration will be 1 year.

STUDY OVERVIEW Appropriate patients with DDDRP pacemakers with an AF burden of 1-50% detected on pacemaker holters will be identified from the pacing clinic list and the Cardiology Outpatient Department at the Eastbourne District General Hospital. They will be invited to take part after a verbal explanation of the study has been given. If agreement is obtained each patient will be given the Patient Information Sheet and allowed time to consider their participation in the study and to ask relevant questions. If they are still in agreement they will be asked to sign the Patient Consent Form.

Initially, all patients will have all baseline parameters assessed. All patients will stop taking their anti-arrhythmic drugs for a period of one week. Patients will then have a three month course of either dronedarone or placebo according to randomisation in a double blinded fashion. Randomisation will be performed by use of random number tables. At three months data will be collected from patient questionnaires and pacemaker Holter.

There will be a one week washout period at this time. Patients will then cross-over to dronedarone or placebo for a three month period. Data from patient questionnaires and pacemaker Holters will be collected at three months after cross-over.

Patients will then undergo a further week washout period before re-initiating their original anti-arrhythmic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal atrial fibrillation (AF burden 1-50% as defined by DDDRP PPM) during the 3 months prior to induction to the study.
* Patients who have had DDDRP pacemaker implanted for a primary or secondary indication.
* Patients must be on warfarin.
* Patients must be over 18 years old.
* Patients give informed consent form prior to participating in this study.

Exclusion Criteria:

* Current or previous treatment with amiodarone.
* Patient is suffering with unstable angina in last 1 week.
* Patient has had a myocardial infarction within last 2 months.
* Patient is expecting or has had major cardiac surgery within last 2 months.
* Patient is participating in a conflicting study.
* Patient is mentally incapacitated and cannot consent or comply with follow-up.
* Patient has NYHA class III/ IV heart failure.
* Pregnancy.
* Patient suffers with other cardiac rhythm disorders.
* Recent coronary artery intervention or other factors suggesting clinical instability (ECG, clinical or laboratory findings).
* GFR < 30mls/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
To accurately assess, by the use of long term beat to beat pacemaker Holter monitoring, the effect of of dronedarone upon AF burden. | 3 months

SECONDARY OUTCOMES:
To accurately assess the number of AF episodes, AF frequency and average duration of sinus rhythm. | 3 months
To assess differences in patient experience of dronedarone and placebo therapies by means of questionnaires. | 3 months
Quality of life measures - SF-36, visual analogue scores, symptom assessment scores. | 3 months
Comparison of side effects and major adverse cardiac events. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: A N Sulke, MD, Principal Investigator — East Sussex NHS Trust
Locations (1):
- Eastbourne DGH, Eastbourne, East Sussex, United Kingdom